CLINICAL TRIAL: NCT00563875
Title: Laboratory Aspirin Resistance in Coronary Artery Disease Patients With or Without Diabetes Mellitus
Brief Title: Laboratory Aspirin Resistance in Diabetics and Non-Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Steen Dalby Kristensen, Aarhus University Hospital Skejby
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20070180; DDPA-2007-41-1207; DRA-2101-05-0052
Record Dates: First submitted 2007-11-23; First posted 2007-11-26 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Drug Resistance
Keywords: Platelets; Platelet aggregation; Drug resistance; Aspirin; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: acetylsalicylic acid — 75 mg/d for 7 days (healthy volunteers) and continued treatment with 75 mg/d in patients taking daily aspirin.
  Other Names: Hjerdyl (Sandoz)

SUMMARY:
Despite treatment with aspirin a large number of patients suffer a myocardial infarction. It has been speculated that these patients might be "resistant" to aspirin, and studies have indicated that this phenomenon is related to a less favourable prognosis. Furthermore, patients with diabetes mellitus have an increased risk of myocardial infarction and other vascular events and, recently, it has been suggested that diabetics do not respond adequately to aspirin. The purpose of this study is to compare the prevalence of "aspirin resistance" in diabetics and non-diabetics. Furthermore, patients who suffered a myocardial infarction while being treated with aspirin are included. We hypothesize that the prevalence of "aspirin resistance" will be higher among diabetics compared to other patients and to healthy individuals.

DETAILED DESCRIPTION:
A considerable number of patients suffer acute coronary events despite being treated with antiplatelet therapy such as aspirin. Taken together with laboratory findings of a low response to aspirin, the term "aspirin resistance" has been coined. Diabetics have an increased risk of suffering ischemic vascular events and, recently, an increased prevalence of "aspirin resistance" was reported in these patients. The purpose of the present study is to compare the aspirin response in diabetics and non-diabetics in a population with angiogram-verified coronary artery disease. Furthermore, healthy volunteers and patients who suffered a myocardial infarction while being treated with aspirin are included. Eligible patients are identified in the Western Denmark Heart Registry.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic heart disease verified by coronary angiogram (group:"CAD")
* treatment with aspirin 75 mg/d for at least the previous 7 days(groups: "CAD" and "Previous myocardial infarction")
* type II diabetes mellitus (~50% of groups: "CAD" and "Previous myocardial infarction")
* ≥ 1 myocardial infarction more than one year ago while taking daily aspirin ≥ 75 mg/d (group: "Previous myocardial infarction").

Exclusion Criteria:

* treatment with NSAIDs, clopidogrel, ticlopidine, dipyridamole, warfarin or any other drugs known to affect platelet function.
* ischemic vascular event within the previous 12 months
* revascularization (angioplasty or coronary by-pass graft surgery) within the previous 12 months
* intake of NSAIDs within 1 week of myocardial infarction (group: "Previous myocardial infarction").
* platelet count < 120 x 10^9/l
* previous myocardial infarction (group: "CAD").
* not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation | (at least) one hour after aspirin ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Steen D Kristensen, M.D., DMSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Clinical Biochemistry, Centre for Haemophilia and Thrombosis, Aarhus University Hospital Skejby, Aarhus N, Denmark